CLINICAL TRIAL: NCT04757805
Title: Assessment of the Accuracy of the Manual Palpation of Surface Landmarks Versus Ultrasound for Identification of the Correct Intervertebral Space for Spinal Anesthesia in Children Less Than 1 Year of Age
Brief Title: Accuracy of Manual Palpation vs Ultrasound for Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Giorgio Veneziano, Associate Professor of Clinical Anesthesiology and Pain Medicine, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000558
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2022-09-15 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia, Local; Infant Conditions
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spinal anesthesia (Experimental): Infants receiving spinal anesthesia for standard of care procedure
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound to locate the appropriate lumbar interspace to perform spinal anesthesia.

SUMMARY:
Although the current standard for lumbar puncture and spinal anesthesia is the use of manual palpation of surface landmarks to identify the correct interspace, performance of the procedure at too high of a level may increase the incidence of adverse effects. The current study will evaluate the efficacy of ultrasound in identifying the correct intervertebral space for lumbar puncture thereby improving the safety of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 1 year of age scheduled for spinal anesthesia for elective lower abdominal, urologic, or lower extremity surgery at Nationwide Children's Hospital

Exclusion Criteria:

* Parents unwilling for their children to undergo spinal anesthesia for surgery.
* Children with known spinal anomalies including sacral dimple.
* Children with coagulation abnormalities or receiving anticoagulation which precludes the use of spinal anesthesia.
* Children with superficial or deep infections over the spine which precludes the use of spinal anesthesia.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spinal Anesthesia
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Anesthesia
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 7 [5 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50
Height [Median (Inter-Quartile Range); unit: centimeters] | 66.5 [63.5 to 70.7]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 7.8 [6.8 to 9]
American Society of Anesthesiologists (ASA) status [Count of Participants; unit: Participants] — The ASA score is a subjective assessment of a patient's overall health that is based on five classes (I to V):
  I = Patient is a completely healthy fit patient. II = Patient has mild systemic disease. III = Patient has severe systemic disease that is not incapacitating. IV = Patient has incapacitating disease that is a constant threat to life. V = A moribund patient who is not expected to live 24 hours with or without surgery.
  Participants
    ASA I | 29
    ASA II | 18
    ASA III | 3

OUTCOME MEASURES:

1. Primary Outcome: Intended Interspace
Description: The vertebral interspace that the anesthesia provider believes that they had marked & identified by manual palpation
Time Frame: Immediately prior to spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia
Number analyzed (Participants) | 50
Participants
  L2-3 | 1
  L3-4 | 24
  L4-5 | 25

2. Primary Outcome: Actual Interspace of Provider's Mark
Description: The actual vertebral interspace that the anesthesia provider marked & identified, as verified by ultrasound.
Time Frame: Immediately prior to spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia
Number analyzed (Participants) | 50
Participants
  L2-3 | 5
  L3-4 | 24
  L4-5 | 21

3. Secondary Outcome: Level of Conus Medullaris - Sitting
Description: Assessing the level of the conus medullaris by ultrasound in the sitting position.
Time Frame: Immediately prior to spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Anesthesia
Number analyzed (Participants) | 50
Participants
  T12-L1 | 9
  L1-2 | 27
  L2-3 | 9
  L3-4 | 3
  Unable to obtain | 2

4. Secondary Outcome: Time to Mark
Description: The amount of time if took for the anesthesia provider to manually palpate and mark the desired interspace.
Time Frame: Immediately prior to spinal anesthesia
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Spinal Anesthesia
Number analyzed (Participants) | 50
seconds | 25 [14.3 to 32]

5. Secondary Outcome: Time to Conduct Ultrasound
Description: The amount of time it took for the investigator to identify the actual space that the provider marked using ultrasound.
Time Frame: Immediately prior to spinal anesthesia
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Spinal Anesthesia
Number analyzed (Participants) | 50
seconds | 38.5 [29 to 63.8]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Spinal Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT04757805/Prot_SAP_000.pdf